CLINICAL TRIAL: NCT06287125
Title: Renal Assessment for Early Detection of Renal Impairment in Systemic Sclerosis and Systemic Lupus Erythematosus Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Nabil Badr, assistant lecturer, Assiut University
Other Study IDs: Renal assess in SSc and SLE
Record Dates: First submitted 2024-02-20; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Systemic Sclerosis and Systemic Lupus Erythematous
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- systemic sclerosis patients: Adult (aged above 18 years) SSc patients who fulfilled the 2013 European League Against Rheumatism/American College of Rheumatology (EULAR / ACR) for SSC and 1980 ACR criteria.
  -SSc patients will be subjected to 2017 European Scleroderma Trials and Research group (EUSTAR) activity index
  Interventions: Device: Renal multi-parametric MRI, Renal doppler ultrasound, Serum CD147
- systemic lupus erythematosus patients: Adult SLE Patients who fulfilled the 2019 EULAR / ACR classification criteria for systemic lupus erythematosus.
  -SLE patients will be subjected to SLE Disease Activity Score (SLE-DAS).
  Interventions: Device: Renal multi-parametric MRI, Renal doppler ultrasound, Serum CD147
- Healthy controls: Apparently healthy subjects
  Interventions: Device: Renal multi-parametric MRI, Renal doppler ultrasound, Serum CD147

INTERVENTIONS:
Device: Renal multi-parametric MRI, Renal doppler ultrasound, Serum CD147 — Laboratory investigations:
  erythrocyte sedimentation rate (ESR) Serum C-reactive protein (CRP) complete blood picture (CBC) liver function tests (LFT): aspartate transaminase (AST), alanine transaminase (ALT), serum albumin, serum bilirubin.
  kidney function tests (KFT): serum creatinine and blood urea. Estimated glomerular filteration rate (eGFR) by CKD-EPI Creatinine Equation (2021).
  Complete urine analysis for: proteinuria, urinary casts (hyaline, granular), hematuria (RBCs/ high power field), pyuria (WBCs/ high power field).
  24 hour protein in urine and Creatinine clearance. Complement 3and 4(C3,C4). Immunological investigations : Antinuclear antibody (ANA) and Anti-double stranded DNA (ds-DNA).
  Serum CD147
  Radiological investigations:
  * Chest X-ray
  * Renal Doppler
  * Multi-parametric MRI

SUMMARY:
* Evaluate renal resistive index in SSc and SLE patients for early detection of renal impairment.
* Evaluate renal multi-parametric MRI in SSc and SLE patients for early detection of renal impairment.
* Measure the serum levels of CD147 in SSc and SLE patients and its correlation with renal impairment.
* Correlation between detected markers and other assessment tools.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is an autoimmune disease characterized by endothelial dysfunction, collagen deposition, and fibrosis in the skin and internal organs. Systemic lupus erythematosus (SLE) is a complex, multi-organ autoimmune disease. The presence of autoantibodies and circulating immune complexes can cause vasculitis and damage the endothelial cells, leading to multiple organ dysfunctions. Renal involvement in SSc, ranges from urinary abnormalities, reduction of glomerular filtration rate (GFR), and high resistive indices, to scleroderma renal crisis (SRC). Subclinical renal vasculopathy is characterized by progressive increase of intrarenal stiffness and reduction of parenchymal thickness due to post ischemic fibrosis secondary to the renal Raynaud phenomenon.Conversely, in SLE-related kidney manifestations, renal damage results from glomerular involve-ment secondary to immune-complex acti¬vation. Cluster of differentiation 147 (CD147) is, also named extracellular matrix metalloproteinase inducer (EMMPRIN), a transmembrane glycoprotein in the immunoglobulin superfamily that is widely expressed on the surface membrane of various cells. Higher levels of soluble CD147 were found in SSc patients compared to healthy controls and higher levels in SSc patients with scleroderma renal crisis (SRC). Suggesting that CD147 could be a useful tool for identifying SRC risk. In patients with active SLE, CD147 is overexpressed on CD3 T lymphocytes. Renal resistive index (RRI) is a useful non-invasive technique for evaluation of renal disease activity in SLE patients. It can differentiate between patients with active lupus nephritis (LN) and inactive LN. RRI was higher in SSc patients than other autoimmune diseases since subclinical renal vasculopathy is the main pathogenic mecha¬nism of all SSc renal manifestations.Multiparametric renal Magnetic Resonance Imaging (MRI) shows great promise as a non-invasive method to assess kidney structure and function without exposure to radiation or gadolinium contrast agents. In MRI microstructural changes of lupus nephritis kidney such as inflammatory cell infiltration or fibrosis could influence water molecular movement or diffusion, which indicates that diffusion-weigted imaging (DWI) may become a valuable tool in diagnosis of LN. However in systemic sclerosis there is decline of renal blood flow values that indicate microvascular pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (aged above 18 years) SSc patients who fulfilled the 2013 European League Against Rheumatism/American College of Rheumatology (EULAR / ACR) for SSC [13] and 1980 ACR criteria [14].
2. Adult SLE Patients who fulfilled the 2019 EULAR / ACR classification criteria for systemic lupus erythematosus [15]

Exclusion Criteria:

1. Individuals with other autoimmune diseases.
2. Smoking.
3. Infections as chest infection, hepatitis C, hepatitis B and HIV infection.
4. Tumors as hepatocellular carcinoma.
5. Hypertension, diabetes, heart failure, hepatic diseases, chronic renal failure, intrarenal arteriovenous fistula, obstructive nephropathy and urinary tract obstruction.
6. Contraindication for MRI as implanted metallic devices.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include adult SSc and SLE patients consecutively presented at the rheumatology, rehabilitation and physical medicine department, Assiut university hospital from both inpatient department and outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate serum levels of CD147 in SSc and SLE patients | One year
  Its correlation with renal impairment
Evaluate renal resistive index in SSC and SLE patients | One year
  It's correlation with renal impairment
Evaluate Multiparametric MRI in SSC and SLE | One year
  It's correlation with renal impairment

SECONDARY OUTCOMES:
Utility of CD 147 in ssc and SLE patients | One year
  for early detection of renal impairment inandSLE patients
Utility of renal resistive index in SSC and SLE patients | One year
  For early detection of renal impairment
Utility of Multiparametric MRI in SSC and SLE | One year
  For early detection of renal impairment

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Ahmed Fathi, Prof., Study Director — Assiut University; Marwa Mahmoud Abdelaziz, Prof., Study Director — Assiut University

REFERENCES:
- [Background] Rosato E, Gigante A, Barbano B, Gasperini ML, Cianci R, Muscaritoli M. Prognostic Factors of Renal Involvement in Systemic Sclerosis. Kidney Blood Press Res. 2018;43(3):682-689. doi: 10.1159/000489740. Epub 2018 May 10. PMID 29763902
- [Background] Zhao T, Lin FA, Chen HP. Pattern of Nailfold Capillaroscopy in Patients With Systemic Lupus Erythematosus. Arch Rheumatol. 2020 Apr 20;35(4):568-574. doi: 10.46497/ArchRheumatol.2020.7763. eCollection 2020 Dec. PMID 33758813
- [Background] Gigante A, Barbano B, Gasperini ML, Zingaretti V, Cianci R, Rosato E. Renal Parenchymal Thickness in Patients with Systemic Sclerosis Is Related to Intrarenal Hemodynamic Variables and Raynaud Renal Phenomenon. J Rheumatol. 2020 Apr;47(4):567-571. doi: 10.3899/jrheum.190165. Epub 2019 Jun 15. PMID 31203218
- [Background] Pellicano C, Vaiarello V, Colalillo A, Gigante A, Iannazzo F, Rosato E. Role of kinurenic acid in the systemic sclerosis renal involvement. Clin Exp Med. 2023 Sep;23(5):1713-1719. doi: 10.1007/s10238-022-00962-6. Epub 2022 Nov 27. PMID 36436115
- [Background] Anders HJ, Fogo AB. Immunopathology of lupus nephritis. Semin Immunopathol. 2014 Jul;36(4):443-59. doi: 10.1007/s00281-013-0413-5. Epub 2014 Jan 9. PMID 24402709
- [Background] Muramatsu T. Basigin: a multifunctional membrane protein with an emerging role in infections by malaria parasites. Expert Opin Ther Targets. 2012 Oct;16(10):999-1011. doi: 10.1517/14728222.2012.711818. Epub 2012 Aug 11. PMID 22880881
- [Background] Yanaba K, Asano Y, Tada Y, Sugaya M, Kadono T, Hamaguchi Y, Sato S. Increased serum soluble CD147 levels in patients with systemic sclerosis: association with scleroderma renal crisis. Clin Rheumatol. 2012 May;31(5):835-9. doi: 10.1007/s10067-012-1949-9. PMID 22298186
- [Background] Pistol G, Matache C, Calugaru A, Stavaru C, Tanaseanu S, Ionescu R, Dumitrache S, Stefanescu M. Roles of CD147 on T lymphocytes activation and MMP-9 secretion in systemic lupus erythematosus. J Cell Mol Med. 2007 Mar-Apr;11(2):339-48. doi: 10.1111/j.1582-4934.2007.00022.x. PMID 17488482
- [Background] Abd Elsamea MH, Badr AN, Talaat EARenal, et al. Arterial resistive index as a noninvasive biomarker of disease activity in lupus nephritis patients. Egypt Rheumatologist 2022; 44(3):239-244
- [Background] Rosato E, Navarini L, Gigante A, Cianci R, Margiotta D, Barbano B, Afeltra A. Intrarenal arterial stiffness is increased in systemic sclerosis patients with anti-ribonucleic acid polymerase III antibodies. Rheumatology (Oxford). 2017 Jun 1;56(6):1039-1041. doi: 10.1093/rheumatology/kex051. No abstract available. PMID 28340199
- [Background] Francis ST, Selby NM, Taal MW. Magnetic Resonance Imaging to Evaluate Kidney Structure, Function, and Pathology: Moving Toward Clinical Application. Am J Kidney Dis. 2023 Oct;82(4):491-504. doi: 10.1053/j.ajkd.2023.02.007. Epub 2023 May 13. PMID 37187282
- [Background] Zhang S, Lin Y, Ge X, Liu G, Zhang J, Xu S, Wu G, Chen S, Xu J, Suo S. Multiparameter diffusion-weighted imaging for characterizing pathological patterns in lupus nephritis patients: A preliminary study. J Magn Reson Imaging. 2019 Oct;50(4):1075-1084. doi: 10.1002/jmri.26657. Epub 2019 Jan 18. PMID 30659687
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Ellen Csuka M, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American college of rheumatology/European league against rheumatism collaborative initiative. Ann Rheum Dis. 2013 Nov;72(11):1747-55. doi: 10.1136/annrheumdis-2013-204424. PMID 24092682
- [Background] Preliminary criteria for the classification of systemic sclerosis (scleroderma). Subcommittee for scleroderma criteria of the American Rheumatism Association Diagnostic and Therapeutic Criteria Committee. Arthritis Rheum. 1980 May;23(5):581-90. doi: 10.1002/art.1780230510. PMID 7378088
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Systemic Lupus Erythematosus. Arthritis Rheumatol. 2019 Sep;71(9):1400-1412. doi: 10.1002/art.40930. Epub 2019 Aug 6. PMID 31385462
- [Background] Jesus D, Matos A and Henriques C. Detection of changes in SLE disease activity is highly improved with SLE-DAS as compared to SLEDAI: derivation and preliminary validation of the SLE disease activity score (SLE-DAS). Ann Rheum Dis 2018;77:842-3.
- [Background] Valentini G, Iudici M, Walker UA, Jaeger VK, Baron M, Carreira P, Czirjak L, Denton CP, Distler O, Hachulla E, Herrick AL, Kowal-Bielecka O, Pope J, Muller-Ladner U, Riemekasten G, Avouac J, Frerix M, Jordan S, Minier T, Siegert E, Ong VH, Vettori S, Allanore Y. The European Scleroderma Trials and Research group (EUSTAR) task force for the development of revised activity criteria for systemic sclerosis: derivation and validation of a preliminarily revised EUSTAR activity index. Ann Rheum Dis. 2017 Jan;76(1):270-276. doi: 10.1136/annrheumdis-2016-209768. Epub 2016 Sep 12. PMID 27621285